CLINICAL TRIAL: NCT01052311
Title: The Impact of Tredaptive (ER Niacin/Laropiprant) Compared to Placebo on Brachial Artery Endothelial Function in Patients With Stable Coronary Artery Disease on Statin Therapy
Brief Title: The Impact of Tredaptive on Flow-Mediated Dilation in Cardiac Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The sponsor decided to withdraw study drug from market
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-09-7418-MS-CTIL
Record Dates: First submitted 2010-01-16; First posted 2010-01-20 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Disease; Dyslipidemia
Keywords: Coronary artery disease; Endothelial function; Platelet function; Statins; Niacin
MeSH Terms: conditions — Coronary Artery Disease; Dyslipidemias | interventions — MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo pills once daily
  Interventions: Drug: Placebo
- Active treatment (Active Comparator): Laropiprant (LRP; Merck & Co., Inc, Whitehouse Station, NJ, USA) is a potent, once-daily, highly selective PGD2-receptor (DP1) antagonist. A combination tablet containing 1 g of extended-release niacin and 20 mg of laropiprant (ERN/LRPT) = tredaptive once daily from day 1 to 30. From day 31 to day 90 2 g of extended-release niacin and 20 mg of laropiprant once daily.
  Interventions: Drug: Tredaptive (1 g extended release niacin+ 20 mg laropiprant); Drug: Tredaptive

INTERVENTIONS:
Drug: Tredaptive (1 g extended release niacin+ 20 mg laropiprant) — Laropiprant (LRP; Merck & Co., Inc, Whitehouse Station, NJ, USA) is a potent, once-daily, highly selective PGD2-receptor (DP1) antagonist. A combination tablet containing 1 g of extended-release niacin and 20 mg of laropiprant (ERN/LRPT) once daily for the first 30 days. from day 31 to 90 it will be 2 g of extended-release niacin and 20 mg laropiprant once daily.
  Other Names: Active treatment
  Arms: Active treatment
Drug: Placebo — Placebo tablets once daily
  Arms: Placebo
Drug: Tredaptive — Tredaptive 1 g [Laropiprant 20 mg(LRP; Merck & Co., Inc, Whitehouse Station, NJ, USA) and 1 g of extended-release niacin]from day 1 to 30 once daily. From day 31 to 90, the same but 2 g instead of 1 g of extended-release niacin.
  Other Names: Tedaptive
  Arms: Active treatment

SUMMARY:
Laropiprant (LRP; Merck & Co., Inc, Whitehouse Station, NJ, USA) is a potent, once-daily, highly selective PGD2-receptor (DP1) antagonist. A combination tablet containing 1 g of extended-release niacin and 20 mg of laropiprant (ERN/LRPT) offers improved tolerability, supporting a simplified 1-2 g dosing paradigm and improved adherence. Statins and niacin improve endothelial function in cardiac patients, however, there is no data yet regarding the additive effects of raising HDL-C by ERN/LRPT and statins on endothelial function in cardiac patients. Thus the aim of the present study is to evaluate the impact of 3 months' administration of ERN/LRPT compared to placebo added to statins on endothelial function, assessed by brachial artery vasoreactivity in stable cardiac patients.

DETAILED DESCRIPTION:
Endothelial dysfunction reflects a vascular phenotype prone to atherogenesis and may therefore serve as a marker of an inherent atherosclerotic risk. In line with this hypothesis, dysfunction of either the coronary or peripheral vascular endothelium was shown to constitute an independent predictor of cardiovascular events, providing valuable prognostic information additional to that derived from conventional risk factor assessment. Interventions, such as risk factor modification and treatment with various drugs, including statins and niacin, may improve endothelial function leading potentially to improve prognosis.

Research over the past years has identified numerous beneficial effects of high-density lipoprotein (HDL) beyond this property. These include, but not limited to, improvement of endothelial function, anti-inflammatory, anti-thrombotic, antioxidative effects and the stimulation of endothelial regeneration. Consequently, therapeutic elevation of HDL is among the primary goals of treatment of patients with coronary artery disease (CAD). Laropiprant (LRP; Merck & Co., Inc, Whitehouse Station, NJ, USA) is a potent, once-daily, highly selective PGD2-receptor (DP1) antagonist. A combination tablet containing 1 g of extended-release niacin and 20 mg of laropiprant (ERN/LRPT) offers improved tolerability, supporting a simplified 1-2 g dosing paradigm and improved adherence. Statins and niacin improve endothelial function in CAD patients, however, there is no data yet regarding the additive effects of raising HDL-C by ERN/LRPT and statins on endothelial function in CAD patients. Thus the aim of the present study is to evaluate the impact of 3 months' administration of ERN/LRPT compared to placebo added to statins on endothelial function, assessed by brachial artery vasoreactivity, and platelet function in stable CAD patients .

ELIGIBILITY:
Inclusion criteria:

1. Male or female ≥ 18 years; signed informed consent
2. Outpatient CAD patients on statin therapy.
3. HDL-C < 40 mg/dL in males and < 50 mg/dL in females.
4. Left ventricular (LV) systolic dysfunction ≥ 40% measured within the past 6 months.
5. No changes in cardiac medications during 2 weeks prior to enrollment.

Exclusion criteria:

1. Presence of transplanted tissue or organ or LVAD
2. AICD or CRT or CRTD patients.
3. Acute MI, CABG, PCI within past 3 months.
4. Congestive heart failure (CHF) ≥ NYHA 2.
5. Ejection fraction < 40% measured within the past 6 months.
6. Malignancy.
7. Active myocarditis, or cardiomyopathy.
8. HIV infection or immunodeficiency state.
9. Chronic viral infection.
10. Acute systemic infection requiring antibiotics.
11. Chronic diarrhea or malabsorption.
12. Statin therapy initiation ≤ 3 months.
13. Diabetes mellitus type 1.
14. Diabetes mellitus type 2 with HbA1C > 7%
15. Low-density lipoprotein cholesterol (LDL-C) > 100 mg/dL.
16. Not on statin therapy.
17. Liver function tests (LFT) ≥ x 3 upper limit of normal (ULN) or creatinine kinase (CPK) ≥ x 10 ULN.
18. Hypo/hyper thyroidism.
19. Liver dysfunction.
20. Renal failure with serum creatinine ≥ 2 mg/dL.
21. Alcohol or drug abuse.
22. Refuse to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of 3 months' administration of ERN/LRPT compared to placebo added to statins on endothelial function, assessed by brachial artery vasoreactivity in stable CAD patients. | 3 months

SECONDARY OUTCOMES:
To evaluate the impact of 3 months' administration of ERN/LRPT compared to placebo added to statins on platelet function in stable CAD patients. | 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shechter, MD, MA, Principal Investigator — Leviev Heart Center, Sheba Medical Center; Shlomi Matetzky, MD, Study Director — Leviev Heart Center, Sheba Medical Center
Locations (1):
- Leviev Heart Center, Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No